CLINICAL TRIAL: NCT03163732
Title: A Multicentric, Prospective Cohort Study Aiming to Evaluate the Added Value of a Large Molecular Profiling Panel (Panel FoundationOne) Versus a Limited Molecular Profiling Panel (Panel CONTROL) in Advanced Solid Tumors.
Brief Title: Evaluation of the Added Value of a Large Molecular Profiling Panel Versus a Limited Molecular Profiling Panel in Advanced Solid Tumors.
Acronym: PROFILER 02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ET16-115
Record Dates: First submitted 2017-05-17; First posted 2017-05-23 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-03

CONDITIONS: Advanced Solid Tumor
Keywords: Solid tumor; Advanced tumor; Profiling panel
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: * Arm A: Tumor-based genomics according to the 324 cancer-related genes Next Generation Sequencing (NGS) panel from Foundation One (FOne panel).
  * Arm B: Tumor-based genomics according to the 87 cancer-related genes NGS panel performed at Centre Leon Berard "Unité de Caractérisation Tumorale" (CONTROL panel).
  Both panels will be performed concomitantly for all patients using the same patient tumor specimen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Large molecular profiling panel (Other): This panel is FOne Panel with a 324 cancer-related gene.
  Interventions: Genetic: Blood and tumor samples
- Limited molecular profiling panel (Other): This panel is CONTROL Panel with a 87 cancer-related gene.
  Interventions: Genetic: Blood and tumor samples

INTERVENTIONS:
Genetic: Blood and tumor samples — Evaluation of the added value of a large molecular profiling panel versus a limited molecular profiling panel
  Other Names: Evaluation of the added value of a molecular profiling panel

SUMMARY:
The PROFILER 02 program is a multicenter, randomized, prospective cohort study aiming to compare the clinical relevance of a large Next-generation sequencing (NGS) panel (FondationOne or FOne panel) versus a limited NGS panel (CONTROL or CTL panel) in patients with advanced solid tumors.

This study will allow adapting the therapeutic management of these patients, if needed, by giving them recommended therapies (commercialized or in ongoing clinical trials), based on the recommendations of the Molecular Tumor Board (MTB).

DETAILED DESCRIPTION:
The genetic and immunologic profile of the tumor will be determined from archival or fresh collected tumor sample.

For each patient, the tumor genomics data will be reviewed, at time of documented progressive disease, independently by a dedicated MTB to make a recommendation of therapy for a given patient based on its molecular profile. First, the genomics data issued from the panel defined by the randomization will be reviewed and recommended therapy resulting from randomization will be revealed to the Investigator. If a recommended therapy can be identified, this therapy will be recommended.

If none recommended therapy can be identified, the 2nd panel performed will then be reviewed.

In case of confirmed clinical or radiological progression (at Investigator's discretion) and/or unacceptable toxicity as per Investigator judgment during the line of therapy recommended by the MTB, the results of the second panel will be reviewed by MTB. Based on all genomics data available (i.e. randomized and 2nd panels), the MTB will recommend other treatment options. All results will be disclosed to Investigator in order to offer other treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged ≥ 18 years at time of inform consent signature.
* Currently treated by a first or a second line of chemotherapy for their advanced cancer (local relapse or metastatic; Immunotherapies, Endocrine therapies and Targeted therapies are not considered as a line of chemotherapy).
* Histologically confirmed diagnosis of advanced (local relapse or metastatic), incurable solid tumors from any histological types (except those listed in exclusion criteria 3).
* I4. Availability of an adequate tumor sample to be sent imperatively to the CLB within 15 days after ICF signature by order of preference either (i1) a tumor archival FFPE block not older than 3 months prior to ICF signature or if not available :(ii2) a dedicated biopsy from one accessible lesion visible by medical imaging and accessible to percutaneous sampling with a diameter of at least 10 mm or if not feasible (3) an archival tumor sample (primary tumor or metastatic lesion) not older than 3 years at time of ICF signature. Quality (at least 20-30% of tumor cells) and quantity (sample size surface area > 5mm2 and > 90um depth) of the tumor sample have to be confirmed mandatorily within 7 days by a central pathological review before confirmation of inclusion.
* Patient's disease which is not susceptible to progress during the next 45 days following the ICF signature.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-1.
* Adequate organ and marrow function based on a medical records (within 21 days before randomization) as defined below :

  * Hemoglobin ≥ 9.0 g/dL
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Platelets ≥ 100 x 109/L
  * Lymphocyte count ≥ 1 x 109/L
  * Serum creatinine CL > 50 mL/min per 1.73m2 using MDRD or CKD-EPI
  * AST and ALT ≤ 2.5 Upper Limit Normal (ULN) (up to 5 ULN may be tolerated in case of liver metastases)
  * Serum bilirubin ≤ 1. 5 ULN (in the absence of Gilbert's syndrome).
* Patient should understand, sign, and date the written ICF prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol.
* Patient must be covered by a medical insurance.

Exclusion Criteria:

* Inability to take oral medication or significant nausea and vomiting, malabsorption, external biliary shunt, or significant bowel resection that would preclude adequate absorption of oral medication.
* Any clinically significant and/or uncontrolled medical disease that could compromise the patient's ability to tolerate an anti-cancer treatment and its procedures (these conditions include but are not limited to severely impaired lung function, active gastrointestinal tract ulceration, acute or chronic uncontrolled liver disease/or severe renal disease, uncontrolled diabetes, history of HIV infection/or active viral infection (HBV, HCV), history of organ allograft or patient taking immunosuppressive treatment).
* Patient with the following advanced cancers :

  * Cancer bearing one of the oncogenic driver mutation: Colorectal cancer : KRAS, NRAS, HRAS and BRAF/Lung cancer: ALK, EGFR, ROS or MET/Breast cancers : RH+ and/or HER2+
  * High-grade serous ovarian cancers platinum-sensitive,
  * Liposarcoma.
  * Melanoma: BRAF
* Patient with non assessable tumor sample.
* Patient already included in this study for a type of cancer, can't be included a second time for the same cancer or for any other type of cancer.
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Compare the proportion of patients for whom a genomically identified recommended therapy could be initiated using the large NGS panel from FoundationOne versus the limited CONTROL panel. | 28 months

SECONDARY OUTCOMES:
Compare in the 2 randomization arms the number of patients with at least one actionable alteration. | 28 months
Compare in the 2 randomization arms the proportion of patients for which a genomically identified recommended therapy is effectively initiated. | 28 months
Describe in both arms the number of patients for whom a genomically identified recommended therapy was available but not initiated. | 28 months
Evaluate proportion of patients who could have been initiated a recommended therapy considering only the INCa panel. | 28 months
  Evaluate proportion of patients with at least one actionable alteration and for whom a genomically identified recommended therapy could have been initiated considering only the INCa panel with only 16 cancer-related genes already included in CONTROL panel
Progression-Free Survival (PFS) | 24 months
  Measured from the date of study drugs start to the date of the first objective radiological disease progression using RECIST 1.1 or death.
Overall response Rate (ORR) | 24 months
  the most clinically favorable response recorded from the start of a recommended therapy until the end of treatment, according to RECIST 1.1
Duration of response (DoR) | 24 months
  Calculated from date of first documented objective response (i.e., Complete Response or Partial Response) until date of first documented progression disease (measurements according to RECIST 1.1 criteria).
Patient Quality Of Life | 12 months
  Measured by the questionnaire EuroQoL-5Dimension-3L
Perform a health economic evaluation | 12 months
  A Cost-Effectiveness and a Cost-utility Analyses comparing the two molecular profiling strategies.
Perform a health economic evaluation | 12 months
  A budget impact analysis to estimate the financial consequences of adoption and diffusion of the large FondationOne panel.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Olivier, MD, Principal Investigator — Centre Leon Berard
Locations (15):
- France (15):
  - Institut Bergonié, Bordeaux
  - Centre Jean PERRIN, Clermont-Ferrand
  - Centre Georges François LECLERC, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - Institut Paoli Calmettes, Marseille
  - AP-HM MARSEILLE - Hôpital Nord, Marseille
  - Institut cancer Montpellier - ICM, Montpellier
  - Institut Curie, Paris
  - Hopital Tenon, Paris
  - Centre Eugène Marquis, Rennes
  - ICO site René Gauducheau, Saint-Herblain
  - Institut de Cancérologie Lucien NEUWIRTH, Saint-Priest-en-Jarez
  - Institut Claudius Regaud, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tredan O, Pouessel D, Penel N, Chabaud S, Gomez-Roca C, Delord JP, Pannier D, Brahmi M, Fabbro M, Garcia ME, Larrieu-Ciron D, Ray-Coquard I, Viala M, Italiano A, Tosi D, Cassier P, Dufresne A, Attignon V, Boyault S, Treilleux I, Viari A, Perol D, Blay JY. Broad versus limited gene panels to guide treatment in patients with advanced solid tumors: a randomized controlled trial. Nat Med. 2025 May;31(5):1502-1508. doi: 10.1038/s41591-025-03613-x. Epub 2025 Apr 7. PMID 40195451